CLINICAL TRIAL: NCT06674915
Title: A Single-dose, Open-label, Phase I Study Comparing the Pharmacokinetics, Safety, and Pharmacodynamics of HRS-5965 in Subjects With Mild and Moderate Hepatic Impairment and Normal Hepatic Function
Brief Title: Investigation of Pharmacokinetics,Safety,and Pharmacodynamics of HRS-5965 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-103
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Complement Mediated Primary or Secondary Glomerular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): Subjects with mild hepatic impairment.
  Interventions: Drug: HRS-5965 capsules
- Treatment group B (Experimental): Subjects with moderate hepatic impairment.
  Interventions: Drug: HRS-5965 capsules
- Treatment group C (Experimental): Subjects with normal hepatic function.
  Interventions: Drug: HRS-5965 capsules

INTERVENTIONS:
Drug: HRS-5965 capsules — Oral 50 mg.

SUMMARY:
The study is being conducted to compare the pharmacokinetics, safety, and pharmacodynamics of HRS-5965 in subjects with mild to moderate hepatic impairment and normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study procedures and methods, participate voluntarily and be able to complete the study according to the protocol requirements, and sign the informed consent form (ICF) in writing;
2. Aged 18-70 years old on the date of signing the ICF (including the threshold), both male and female;
3. At the time of screening, male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg; body mass index (BMI): 18~32 kg/m2 (including the threshold);
4. Subjects with childbearing potential must agree to have no plans for childbearing and voluntarily use highly effective contraception with their partner from the time of signing the ICF until 1 month after administration of the test drug, and to avoid sperm/egg donation. Female subjects of childbearing potential must have a negative serum pregnancy test at both screening and baseline and not be breastfeeding.

   For subjects with hepatic impairment, the following inclusion criteria must also be met:
5. Not on medication within 4 weeks prior to screening, or have at least 4 weeks of stable medication for hepatic impairment and/or other co-morbidities requiring long-term treatment;
6. Child-Pugh classification of Class A or B.

   For subjects with normal hepatic function, the following inclusion criteria must also be met:
7. The demographic means of subjects in the normal liver function group (Group C) at screening must meet the following matching criteria:

   1. Weight matched to the hepatic impairment group (Group A + Group B) with a mean value ± 10 kg;
   2. Age-matched to the hepatic impairment group (Group A + Group B), mean ± 10 years;
   3. Sex-matched to liver impairment group (Group A + Group B), mean value ± 1 case;
8. Normal or abnormal physical examination, 12-ECG, vital signs, chest frontal and lateral radiographs/CT, abdominal ultrasound, and laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function, etc.) in the screening and baseline periods were not clinically significant.

Exclusion Criteria:

1. Allergic to two or more allergens, or in the judgment of the investigator, may be allergic to the study drug or its components;
2. Disease or medical condition that, in the judgment of the investigator, may interfere with the absorption, distribution, metabolism, and excretion of the drug or that may reduce compliance;
3. Prior history of meningococcal infection or a first-degree relative with a history of meningococcal infection;
4. Existing or suspected infection (at the investigator's discretion) within 2 weeks prior to screening, or fever;
5. Severe trauma or undergone surgery within 8 weeks prior to screening, or plan to undergo surgery during the trial period;
6. Participated in a clinical trial of any other drug or medical device within 3 months prior to screening or plan to do so during the study period, or still within 5 half-lives of the drug prior to screening (whichever is longer);
7. Smoked an average of more than 5 cigarettes per day in the 4 weeks, or consumed an average of more than 15 g of alcohol in a day in the 4 weeks prior to screening (15 g of alcohol is equivalent to 450 mL of beer, 150 mL of wine, or 50 mL of low-potency liquor), or a positive breath alcohol test at baseline;
8. History of drug or substance abuse; or a positive urine drug test at screening;
9. Donated or lost ≥ 400 mL of blood within 8 weeks, or received a blood transfusion within 12 weeks prior to screening;
10. Malignant tumor, or history of a malignant tumor within 5 years prior to screening (except for primary hepatocellular carcinoma treated with radical surgery without recurrence within 2 years, non-melanoma of the skin for which treatment has been administered without signs of recurrence, and resected cervical intraepithelial neoplasia);
11. Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg at screening;
12. QTcF (males) > 450 ms and a QTcF (females) > 470 ms at screening, or other 12-ECG abnormalities judged by the investigator to be clinically significant or unsuitable for participation;
13. Glomerular filtration rate (eGFR) < 75 mL/min/1.73m2 calculated using the Chronic Kidney Disease Epidemiology Collaborative Study Group (CKD-EPI) formula;
14. Difficulty in swallowing, collecting blood intravenously, or physically unable to tolerate blood collection, or not expected to complete the entire trial follow-up;
15. Vaccinated within 2 weeks prior to dosing or plan to receive the vaccine during the study and within 1 month after dosing;
16. Pre-existing recurrent oral ulcers;
17. Any physical or psychological disease or condition that, in the judgment of the investigator, is likely to increase the risk of the trial, interfere with compliance with the protocol and ability to complete the trial.

    Additional exclusion criteria for subjects with hepatic impairment (excluded if 1 of these criteria is met):
18. History of liver transplantation;
19. Liver failure, or cirrhosis with combination of hepatic encephalopathy, hepatocellular carcinoma, ruptured variceal hemorrhage of the esophagogastric fundus vein, and other complications that, in the judgment of the investigator, make the subject unsuitable for participation in the study;
20. History of any serious disease other than the primary disease of the liver itself, or a history of and/or abnormal clinically significant clinical laboratory tests that, in the opinion of the investigator, may affect the results of the test, including, but not limited to, a history of circulatory, endocrine, neurological, gastrointestinal, urologic, or hematologic, immunologic, psychiatric, and metabolic disorders;
21. Positive Human Immunodeficiency Virus (HIV) antigen/antibody screen; if syphilis spirochete antibody is positive, additional tolulized red unheated serum test (TRUST) is required, and exclusion is required if TRUST is positive at the same time; if Hepatitis B Surface Antigen (HBsAg) is positive, additional Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Quantitative Test is required, and if Hepatitis C Virus If hepatitis C virus (HCV) antibody (Anti-HCV) is positive, additional quantitative hepatitis C virus (HCV) ribonucleic acid (RNA) testing is required, and exclusion will be determined by the investigator based on the quantitative results;
22. Alpha-fetoprotein > 20 ng/mL; hemoglobin (Hb) ≤ 70 g/L; alanine aminotransferase (ALT) or mentholatum aminotransferase (AST) ≥ 5 times the upper limit of normal (ULN);
23. On systemic hormones (except subjects on stable use of ≤ 5 mg/day of prednisone or equivalent doses of glucocorticoids) or other immunosuppressive agents within 4 weeks prior to screening, or more than 4 weeks from their last immunosuppressive therapy at screening but are still within the drug's efficacy period (as assessed by the investigator);
24. On herbal medications within 4 weeks prior to screening;
25. On albumin within 14 days prior to screening.

    Additional exclusion criteria for subjects with normal hepatic function (excluded if 1 of these criteria is met):
26. Pre-existing serious primary diseases of vital organs, including but not limited to gastrointestinal, respiratory, renal, hepatic, neurological, hematological, endocrine, oncological, immunological, psychiatric, or cardiovascular diseases;
27. Positive for any of the HBsAg, Anti-HCV, HIV antigen/antibody, or syphilis spirochete antibody tests;
28. On any medication (including prescription drugs, over-the-counter medications, herbal medicines, proprietary Chinese medicines and dietary supplements, etc.) within 4 weeks prior to screening; or within 5 half-lives of the medication at the time of screening (whichever is longer).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Cmax | Post-dose at day 1 to day 9.
  The maximum plasma concentration.
AUClast | Post-dose at day 1 to day 9.
  Area under the concentration curve from time 0 to the last quantifiable concentration.
AUCinf | Post-dose at day 1 to day 9.
  Area under the concentration curve from time 0 to extrapolated infinite time.

SECONDARY OUTCOMES:
Tmax | Post-dose at day 1 to day 9.
  Time to maximum plasma concentration.
t1/2 | Post-dose at day 1 to day 9.
  Terminal half-life.
CL/F | Post-dose at day 1 to day 9.
  Apparent clearance.
Vz/F | Post-dose at day 1 to day 9.
  Apparent volume of distribution.
Incidence and severity of adverse events | Screening period up to day 9.
Change from baseline of alternative pathway activity | Post-dose at day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided